CLINICAL TRIAL: NCT07012473
Title: The Effect of Nutrition Education on the Consumption of Green Leafy Vegetables and Legumes and the Potential Impact on Nutrition in the Accra Metropolitan Area, Ghana
Brief Title: Effect of Nutrition Education on Vegetable and Legume Intake Among Households in Accra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ghana (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Patience Atitsogbey, Principal Investigator, University of Ghana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CBAS 004/21-22
Record Dates: First submitted 2025-05-24; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiency Anemia
Keywords: Nutrition education; Green leafy vegetables; Legumes; haemoglobin levels; iron-bioaccessibity; parents-child pair; Ghana
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: There will be two groups but only one group ( the interventiongroup) will receive the intervention while the second group will not receive the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Intervention Group: Will receive Nutrition Education Intervention for 6 months
  Interventions: Behavioral: Nutrition education on green leafy vegetables and legumes
- Control Group (No Intervention): Control Group: This group will not be given any form of Nutrition Education from the researcher for 6 months period

INTERVENTIONS:
Behavioral: Nutrition education on green leafy vegetables and legumes — The nutrition education intervention will be based on the Theory of Reasoned Action, Social Cognitive Theory, and the Health Belief Model to influence key behaviour change factors such as knowledge, attitudes, practices, and beliefs. Educational materials will include stickers featuring indigenous green leafy vegetables, legumes, and vitamin C-rich fruits, with information on their benefits, storage, preparation, and the importance of combining them for enhanced iron absorption. Other materials include videos, messages, and affirmative words on iron deficiency and its prevention. The intervention will be delivered to selected households in the intervention community through biweekly meetings and phone calls over six months. The control community will not receive any intervention from the researcher.
  Arms: Intervention Group

SUMMARY:
The main purpose of this observational study is to determine the effect of nutrition education on the knowledge and behaviour of households towards the consumption of green leafy vegetables, legumes and vitamin C-rich fruits and its influence on haemoglobin levels of (households) mothers, fathers and children. The questions it aimed to answer are:

* What is the effect of nutrition education on knowledge, attitude and practice towards the consumption of green leafy vegetables and legumes among households in Ayawso Central Municipality?
* What are the consumption patterns of green leafy vegetables, legumes and vitamin C -rich fruits among households in Ayawso Central Municipality?
* What is the iron, β-carotene, vitamin C and antinutritional contents of the commonly consumed green leafy vegetables and legumes in Ayawso Central Municipality?
* Is iron bioaccessible in the commonly consumed green leafy vegetables and legumes in Ayawso Central Municipality?
* What is the haemoglobin level of participants at baseline and end line in Ayawso Central Municipality?

The study will address knowledge, attitude and the low intake of these nutrient-rich foods and the high prevalence of iron deficiency anaemia/ anaemia among women, children and men through nutrition education and also examine the iron content and iron bioaccessibility in the indigenous green leafy vegetables and legumes that participants consume.

Participants are aware of indigenous green leafy vegetables, legumes and vitamin C-rich fruits in their environment; however, they do not consume them frequently. They will answer questions on knowledge, attitude and practices towards these foods during the six months study and have their haemoglobin levels determine.

DETAILED DESCRIPTION:
Background Green leafy vegetables and legumes are important sources of essential nutrients such as dietary fibre, protein, vitamins, minerals (including iron, zinc, and calcium) and phytochemicals required for growth and development. Despite their nutritional benefits, the consumption of these foods remains low in many parts of the world, including Ghana. A significant barrier to the low consumption of these vital foods is inadequate knowledge and awareness regarding their nutrient content and health importance.

Recent evidence suggests that consumption of green leafy vegetables and legumes has the potential to improve iron status and alleviate iron deficiency anaemia and hidden hunger among women and children. Iron is an essential micronutrient for human health throughout the life cycle. Its deficiency results in iron deficiency anaemia (IDA) which constitutes a major public health problem worldwide, affecting women of reproductive age and children but mostly predominant in the developing.

Globally, about 614 million women of reproductive age (15-49 years) and 280 million children are anaemic, with iron deficiency being a principal cause. However, in Africa, the highest prevalence of iron deficiency anaemia cases are found in Central and West Africa where about 71% of children under five years are anaemic.

Problem statement Inadequate consumption of green leafy vegetables and legumes is prevalent among households in Accra, Ghana, leading to a high prevalence of diet-related diseases and deficiencies such as anaemia, iron and vitamin A deficiency, hypertension, diabetes, overweight and obesity. The World Health Organization recommended the intake of 400g (5 servings; 80g per serving) of vegetables and 160g of legumes per day . However, according to recent studies, majority of Ghanaians do not meet the recommended intake of vegetables and legumes, and this can be attributed to insufficient nutrition education. Inadequate nutrition education about the health benefits of foods containing essential nutrients results in their low consumption.

In Ghana, the prevalence of anaemia among women of reproductive age (15-49 years) remains a significant public health concern. Specifically, about 51% of pregnant women, 40% of non-pregnant women and 49% of children under-five years were reported to be anaemic in 2022 .This high prevalence is notably attributed to iron deficiency, mainly resulting from inadequate dietary consumption.

Nutrition education can play a crucial role in promoting healthy dietary behaviours, including the consumption of green leafy vegetables and legumes. Globally, several studies have been conducted to investigate the impact of nutrition education on dietary behaviours in various settings. For example, a study in 2019 and 2016 showed that nutrition education interventions in the USA significantly increased the consumption of vegetables and legumes among adolescents and households. Similarly, a study in India found that nutrition education was effective in promoting the consumption of green leafy vegetables and legumes among households and similar results were observed among Nepalese school children.

However, nutrition education intervention approach has not been explored to promote healthy dietary behaviour among households in the Accra Metropolitan Area. Therefore, it is imperative to adapt nutrition education intervention to promote the consumption of green leafy vegetables and legumes among poor urban households in Accra characterized by low consumption of these foods and a high prevalence of anaemia and iron deficiency. This may lead to improved consumption patterns of these foods which may translate into improved haemoglobin levels among participants.

Specific Objectives

The specific objective of this study are:

1. To determine the effect of nutrition education on knowledge, attitude, and practice of households on green leafy vegetables and legumes consumption.
2. To determine the consumption patterns of green leafy vegetables, legumes, and vitamin C fruits among the households
3. To determine the effect of nutrition education on the haemoglobin level of study participants
4. To determine the chemical composition (moisture, iron, β-carotene and vitamin C and antinutrients- phytate and tannins contents) in the commonly consumed green leafy vegetables and legumes
5. To determine iron bioaccessibility in the commonly consumed green leafy vegetables and legumes

Methodology:

The study was in the following phases:

1. Key informant interview and Focus Group Discussion
2. Intervention study
3. Laboratory investigations on selected green leafy vegetables and legumes

   Key Informant Interview Key Informant interviews (KII) will be carried out among seven (7) people: two (2) elderly men and two elderly women, one community health nurse, one nutrition officer, and one Women in Agriculture Development (WIAD) officer who will be purposively selected. The key informant interview will be used as formative research to understand the background of the study community with regards to cultural practices, green leafy vegetables, legumes, and fruits consumption, food sources, knowledge on iron deficiency anaemia, and anaemia prevention methods employed by community members. A key informant interview (KII) guide will be used to conduct the interview. The information collected will be audiotaped.

   Transcription and Analysis The audio recordings of the key informant interviews will be entrusted to an independent individual for verbatim transcription. The transcripts will then be subjected to a meticulous review carried out by a separate individual. This examination will include attentively listening to the initial voice recordings and verifying them against the transcribed copies. The transcripts will undergo further examination, leading to the creation of a comprehensive codebook. This book will comprise diverse codes accompanied by their definitions, examples of their application, and illustrative instances. After completing the transcription and review stages, the transcripts will be imported into the dedooseTM software, and parent and child codes will be created from the codebook within the dedooseTM software platform. The interpretation of the qualitative data will be based on thematic content analysis.

   Study Area The research will be carried out in two communities within Ayawaso Central Municipal Assembly, located in the Greater Accra Metropolitan Area.

   Sample size determination The estimated sample size calculation will be based on the difference between two independent means (two groups) with the following study parameters in GPower version 3.1.9.7: Alpha: 0.05, Power: 0.80, Effect size: 0.5, N = 102. With a 15% attrition rate added, the total sample size for the study was 117.3, rounded up to 120.

   Sampling of Study Participants A multiple-stage cluster sampling technique will be employed to partition each town into three primary clusters. Within each main cluster, one cluster will be randomly selected using Enumeration Areas (EA), resulting in a total of three clusters per town and six clusters overall for the study. In each selected cluster, the "spinning a bottle" method will be utilized, which involves following a designated path to conduct a systematic sampling of houses. Starting from the first house, every eighth (8th) house will be selected, and this household selection process will be repeated in all the clusters.

   A record of eligible households will be compiled in each selected house. Subsequently, a simple random sampling method involving balloting will be employed to select one eligible family that satisfied the inclusion criteria of the study. To determine the intervention and control towns, one of the towns will be randomly selected as the intervention town, while the second town will serve as the control. Within each town, a total of 60 households that fulfilled the inclusion criteria and are willing to participate in the study will be recruited after signing a consent form. A total of 120 households will be enrolled in the study.

   Household survey data collection. Household data will be collected at three distinct time points: baseline (before the implementation of the intervention), midline (three months after the intervention), and end line (six months after the intervention). Also, the questionnaire will be used to collect information on the household's awareness (only at baseline), knowledge, attitude, and practice with regard to iron, iron-rich foods and iron deficiency anaemia (IDA). Furthermore, a food frequency questionnaire from FAO (2018) will be adapted and used to measure the consumption patterns of indigenous green leafy vegetables, legumes, and vitamin C-rich fruits among participants in the intervention and control group. In addition to the outcome variables, data on the participants' demographic characteristics, including sex, age, occupation, income, educational level, and place of residence, will be collected.

   Biochemical data (Hb and malaria status) collection will involve the use of specific tools and materials. These will include micro cuvettes, lancets, a haemocue device (URIT-12 haemoglobin meter), 70% ethanol, cotton wool, and disposable hand gloves. Blood samples will be obtained by pricking the fingertips of study participants. These samples will be used to determine the haemoglobin levels of households participating in the study within the intervention community. Furthermore, malaria status of households in the intervention community will be assessed using a rapid Diagnostic Test kit (BiolineTM Malaria Ag P.f by Abbot Diagnostics Korea Inc. REF 05FK50). These tests will be conducted at two time points: baseline (0 months) and endline (6 months).

   Data Analyses The household survey data collected in this study will be inputted and analysed using SPSS version 26, a statistical software package. Frequencies and proportions will be used to summarise the categorical data, whereas means and standard deviations will be employed to summarise the continuous variables. All analyses will be considered significant at p < 0.05. Below is the detail of how the various items on the questionnaire will be categorized and scored for the statistical Analysis Knowledge, Attitude and Practices Data on knowledge, attitude, and practice will be analysed using repeated ANOVA to conduct a pairwise comparison across the three data collection points (baseline, midline and endline). A comparison will be made between the intervention and the control group to ascertain whether there existed any difference in the means between the two groups. Covariates such as sources of information (radio, tv, hospitals, family/friends), level of education, ethnicity, and income will be included in the model.
   1. Knowledge The knowledge section comprised questions on recognition of iron-rich foods, iron deficiency anaemia (IDA), signs of iron deficiency anaemia, consequences for pregnant and lactating women and children, causes and strategies for IDA prevention, and foods that enhances or decreases iron absorption. Participants who will indicate that they have knowledge and will be able to select a correct answer or a correct answer plus a correct follow up answer will be assigned a score of one (1) and classified as knowledgeable while those who reported "don't know" will be assigned zero (0) and classified as having no knowledge.
   2. Attitude The section on attitude will comprise questions that measures participants' perceptions of their likelihood of becoming iron deficient.

   Participants will be assigned a score of one (1) if they testify to the following:
   1. They and their children are likely to suffer from iron deficiency anaemia.
   2. IDA is a serious disease.
   3. It is good to cook with iron-rich foods.
   4. They feel confident cooking with iron-rich foods.
   5. They like the taste of meals prepared with iron-rich foods. These groups of participants will be classified as having a good attitude. However, participants who choose not likely, am not sure, not serious, it is difficult, I dislike the taste and not confident will be classified as having a bad attitude and assigned a score of zero (0).

   (c) Practice Several questions on iron-rich foods will be included in the practice section which will evaluate whether participants frequently eat these foods as a whole meal or just a portion of one, and whether they had done so in the week prior to the assessment. Indigenous green leafy vegetables such as cocoyam leaves, jute leaves, water leaves, turkey berries, and legumes such as white beans, red beans, soybeans, and groundnuts known to be common in the communities based on formative research will be included in the questionnaire. Also, animal source foods, such as meat, organs, and both river and sea fish, eggs, and milk, will be also included in this section. The study will also examine whether individuals frequently eat fruits high in vitamin C and how long they cook their green leafy vegetables.

   Furthermore, participants will be asked about their daily tea or coffee consumption and when they drink it if they indicated that they did so. A score of one (1) will be assigned to participants who will answer yes to consuming green leafy vegetables, legumes, and animal source foods. Also, a score of one (1) will be assigned to participants who consume vitamin C-rich fruits. These participants must consume these fruits every day or at least 3-4 times/ 5-6 times per week and tick "No" for tea or coffee or do not consumption immediately before or after meal or during meal. This group of participants will be classified as having good practice. A score of zero (0) will be assigned to a "Yes" to tea or coffee or consumes tea or coffee immediately before or after a meal or during a meal, and "No" to usually consuming green leafy vegetables, legumes, vitamin C rich-fruits or 1-2 times per week and to animal source foods. This group of participants will be classified as having a bad practice.

   Haemoglobin Assessment Haemoglobin levels will assessed in accordance with World Health cut-off points and the standard unit of g/dL. A paired t-test will be employed to investigate the significance of mean differences in haemoglobin levels between the baseline and endline data collected from households within the intervention community. Also, a multivariable test will be performed using a general linear model to investigate the effect of nutrition education on the haemoglobin levels of participants.

   Laboratory Evaluation of Green Leafy Vegetables and Legumes:

   Sampling of Green leafy vegetables and Legumes Sampling point: Findings derived from a formative research carried out in the intervention community revealed that households acquire most of their green leafy vegetables and legumes from two markets, namely Mallam Atta and Agbogbloshie. Consequently, green leafy vegetables and legumes will be sampled within these two markets.

   Stratified Sampling In the two markets, there are specific areas/shades designated for the vending of each food group by the market Queen Mothers and the Municipal Assembly. Green leafy vegetables and legumes will be purchased from sellers who will be in these demarcated areas. To ensure unbiased sampling, the vendors selling various green leafy vegetables and legumes in these specific areas within the two markets will be grouped into strata. Within each stratum, a systematic sampling approach will be employed to select the vegetables. In each market, sampling will begin from the eastern side of the long shades, starting with the second seller from the right side and continued towards the left, from every fifth seller until the entire stratum will be covered, thus ensuring representative sampling. In each market, green leafy vegetables will be sampled from eight sellers and five legume sellers.

   Duplicate samples of the green leafy vegetables and legumes will be purchased at a week interval. The green leafy vegetables that will be acquired from the markets include Xanthosoma sagittifolium (cocoyam leaves), Corchorus olitorius (jute leaves), Solanum macrocarpon (African eggplant), Talinum triangulare (water leaves), Spinacia oleracea (spinach), Taraxacum officinale (dandelion), and Solanum torvum (turkey berry) which is classified as a fruit vegetable. The green leafy vegetables will be identified and verified by a plant and environmental biologist at the Herbarium section of the Department of Plant and Environmental Biology, School of Biological Sciences, University of Ghana. The purchased legumes will include Vigna unguiculata (White beans or cowpea black eye), Vigna angularis (red beans), Vigna subterranea (Bambara beans), Glycine max (Soybeans) and Arachis hypogaea (Peanuts). A crop scientist at the Department of Crop Science, University of Ghana, Legon, will identify the legumes. The procurement of green leafy vegetables and legumes from the markets will take place between 4:00 am to 5:00 am. They were immediately transported on a cold chain to the laboratory of Food Research Institute for subsequent sample preparation.

   Sample preparation The green leafy vegetables will be carefully detached from their stalks, ensuring that only intact and undamaged leaves will be selected for subsequent processing. They will be thoroughly washed under running tap water, followed by a comprehensive rinse using deionized water. The washed samples will be air-dried at room temperature before being finely cut into smaller pieces using sterilized scissors. Approximately 400g of the chopped leafy vegetables will be steamed for a duration of 3 minutes. This steaming process take place on a stainless-steel steamer with 60ml deionized boiling (100 ⁰C) water. The chopped vegetables on the steamer will be covered, allowing them to be cooked by the rising steam. The steamed vegetables will be cooled at room temperature. Once cooled, the steamed samples will be transferred into labelled zip-lock bags for identification purposes and immediately stored in a freezer set to -18 ⁰C for a day. Subsequently, the samples will be transported on a cold chain for freeze-drying.

   Regarding the legumes, approximately 400g of the legume varieties will be soaked in deionized water at room temperature for a duration of 6 hours, following the procedure described by (Nakitto et al., 2015). After soaking, the beans will be drained and rinsed before being boiled with deionized water until they attain a desirable texture characterized by softness without the addition of salt. Once cooked, the legumes will be cooled at room temperature. Subsequently, the legumes, and any remaining cooking liquid from the saucepan will be transferred into labelled zip-lock bags. The bags will be promptly stored in a freezer set at -18 ⁰C for a day and then transported on a cold chain for freeze-drying.

   In the case of peanuts, they will be roasted for a duration of 25 minutes, following which they will be cooled at room temperature. The roasted peanuts will then be transferred into appropriately labelled zip-lock bags and stored in a freezer set to -18 ⁰C for a day and transported on a cold chain for freeze-drying.

   Freeze Drying Procedure The samples will be pre-frozen in a -80 ⁰C freezer for 24 hours, then transferred into a freeze dryer (Supermodulyo, Thermo Scientific) and will be subjected to a drying cycle at a temperature of -35 ⁰C and at a pressure of 25mbar for 72 hours. The dried samples will then be collected and sealed in air-tight zip-lock bags and stored at room temperature for further analysis.

   Milling Procedure The freeze-dried green leafy vegetables and legumes will be milled using a Kenwood dry matter blender and sieved into a fine powder using a stainless-steel mesh with a 0.5ml (500µm) pore size. The flour will be then weighed and transferred into a labelled zip-lock bag and stored at room temperature in the laboratory for further analysis.

   Defatting Procedure of Peanut for Iron Analysis To extract oil from the peanut sample, 30ml of hexane will be added to 5g of the sample contained in a 50ml centrifuge tube. The tube will be then placed on a rotary mixer set at 40rpm for a duration of 3 hours. After the mixing process, the tube will undergo centrifugation at 3000 relative centrifugal force (rcf) for 10 minutes. The resulting clear supernatant will be carefully decanted into a bottle without disturbing the sample.

   This extraction process will be repeated three (3) times, and the duration of shaking will be reduced to 1 hour for each subsequent repetition. In total, four (4) washes will be carried out to ensure thorough extraction. Subsequently, the sample tube will be left loosely capped in a fume cupboard for two days to allow the remaining hexane to evaporate. Next, the sample will be placed in a hot air oven at a temperature of 40 ⁰C for a period of 24 hours and weighed.

   Chemical Composition of Green Leafy Vegetables and Legumes

   Β-Carotene and Vitamin A determination The quantification of β-carotene content in the dried green leafy vegetables and legumes will be assessed through the Spectrophotometric method per the standards specified in ISO BS EN 12823:1-2014. Precisely 5g of the samples will be weighed, and 300mg of Ascorbic acid will be added. This will be followed by adding 15ml of KOH (60%) and 50ml of ethanol to the content in a 250ml flat bottom flask and swirled. The flask will be tightly closed using a stopper and subjected to vigorous shaking. The resultant mixture will be heated to a boiling point while undergoing reflux in a water bath, which will be pre-heated to 90 ⁰C and maintained for 30 minutes. The content of the condenser will be cooled at room temperature, and the saponified solution will be quantitatively transferred into a separating funnel via a series of rinsing using 50ml ethanol, 120ml distilled water, and 150ml of petroleum ether (50ml x3). The extraction obtained will filtered through anhydrous sodium sulphate to remove any possibly suspended drops of water. The extracts will be subjected to evaporation until completely dried, and the dried extracts will be reconstituted with 10ml of petroleum ether. The reconstituted extract will be vortexed and read in the spectrophotometer at the wavelength of 453nM.

   Formula for β- Carotene concentration (mg/100g):

   [Amount of calibration curve(mg) x150x10x100 x F] [100ml x W x V] Where 150 = volume of petroleum ether used 100 = per 100g of sample 10 = volume reconstituted with 10ml ethanol w = weight of sample v = volume of sample (extract) before evaporation F= dilution factor Vitamin A (Retinol Activity Equivalents) The β-carotene values obtained were converted into vitamin A (RAE); assuming 6μg of β-carotene:1μg of retinol

   Vitamin C The content of vitamin C will be quantified by employing the 2,6 dichlorophenolindophenol method with minimal modification. Approximately 1g of the samples will be accurately weighed and placed in a 150ml beaker. Subsequently, 100ml of distilled water will be added to the sample in the beaker. The blend will be left at room temperature for one hour. The resulting supernatant will be separated by filtration into a 150ml conical flask. To the filtrate, 5ml of 20% metaphosphoric acid was added, followed by the addition of 2ml of concentrated acetone. The filtrate containing the sample extract will be then titrated against a solution of 2,6-dichloro indophenol dye. The dye solution (formulated by dissolving 0.05g of the dye in 100ml of distilled water) will be used to fill the burette. The titre value will be carefully recorded for the calculation of the vitamin C content.

   Formular for calculating vitamin C content (mg/100g):

   Mass = titre (raw vitamin C) x mass (pure Ascorbic Acid) x100 titre (pure Ascorbic Acid) x weight of sample

   Iron Content Determination Acid Digest Procedure for ICP-MS Quantitative Iron Analysis The determination of iron content in the samples will be carried out in accordance with the protocol established with minimal modification. A precise amount of 0.05g of milled dried green leafy vegetables and legumes will be weighed into borosilicate tubes that will be washed with acid. Then, 2ml of concentrated nitric acid (HNO3) will be added to the samples, which will be subsequently mixed using a vortex shaker. The tubes will be placed on a pre-heated block with a marble on top to facilitate reflux of the acid. The temperature of the heat block will be gradually increased to 109⁰C and maintained at this temperature for 15 minutes.

   Afterward, the samples will be withdrawn from the heat block and cooled for 15 minutes. To the cooled samples, 1ml of concentrated hydrogen peroxide (H2O2) will be added in increments of 0.25ml, and the mixture will be agitated on a vortex shaker. The samples will be then placed back on the heat block with a marble on top. The temperature of the heat block will be gradually increased to 120⁰C and maintained at this temperature for 2 hours.

   Following this, the samples will be again taken off the heat block and permitted to cool for 15 minutes. Subsequently, 2ml of concentrated nitric acid (HNO3) will be added to the samples, ensuring that the inside of the tube walls is washed to collect any remaining undigested particles. The samples will be again placed on the heat block with a marble and heated at 120⁰C for an additional 2 hours. After cooling for 15 minutes, the samples will be diluted with ultrapure deionized water (UDI) to near the top of the tubes.

   The digested samples will be transferred to 50ml centrifuge tubes, and the digest tubes will be rinsed three (3) times with UDI, and the residual rinsed water will be added into the centrifuge tube. The digested samples will be brought up to a final volume of 40ml. Subsequently, the digested samples will be filtered through a 0.22µm PES Millipore filter into a clean 50ml centrifuge tube.

   The centrifuge tubes will be labelled with the sample name and "10% HNO3" and stored at room temperature. For further analysis, 2ml of the digested sample will be diluted to a final volume of 10ml using UDI, resulting in a 5-fold dilution to produce a matrix with a 2% HNO3 concentration. Elemental analysis will be performed using inductively coupled plasma mass spectrometry or ICP-MS (Thermo-FisherScientific iCAP-Q; Thermo Fisher Scientific).

   Total Iron Concentration (mg/100g) = Cd x V x D W

   Where:

   Cd = iron concentration in the food digest V = extract volume D = dilution factor W = weight of sample used in the digestion procedure

   Antinutrient Determination Phytate Phytate content will be determined in the dried and milled green leafy vegetables and legumes following the method outlined by (Umeobika et al., 2015). Specifically, 0.2g of the samples were weighed into a 250ml conical flask. The sample will be soaked with 50ml of 20% hydrochloric acid (HCl) for a duration of three hours. After the soaking period, the resulting mixture will be filtered into a 250ml beaker.

   To the filtrate, 100ml of distilled water will be added. Successively, 10ml of a 0.3% solution of ammonium thiocyanate will be added to the filtrate. Titration will be performed using a standard solution of iron (III) chloride, which will have a concentration of 0.00195g/ml.

   During titration, a distinctive wine colouration will be expected, indicating the reaction between the phytate and the iron (III) chloride. This colour change will serve as an indicator for the quantification of phytate content in the sample.

   Calculation:

   Phytic acid (mg/100g): Titre ×0.00195× 1.19 ×100 2 Tannins Tannins content will be determined following the methodology described by (Tuli et al., 2016). Approximately 0.2g of the sample will be weighed into a 100ml beaker. To extract the soluble components from the insoluble, 10ml of 70% acetone will be added to the content of the beaker. The resulting mixture will be filtered into a 50ml volumetric flask.

   After filtration, 2ml of 10% anhydrous sodium carbonate solution will be added to the content of the flask. Additionally, 2.5ml of Folin-Ciocalteu reagent will be added. A 70% acetone will be used to top up the content of the flask to the 50ml capacity.

   The prepared mixture will be incubated at room temperature for a duration of 40 minutes. To establish a blank reference, a separate mixture containing all the reagents but excluding the sample will be prepared. Subsequently, the absorbance of the solutions will be determined at a wavelength of 700nm in a UV spectrophotometer. This measurement will allow for the determination of tannin content based on the absorbance values obtained

   Calculation:

   Tannins (mg/100g): Absorbance × Volume Constant Weight 10

   Determination of Iron Bioaccessibility The method that will be employed for determining the bioaccessibility of iron will follow the Simple Bioaccessibility Extraction Test (SBET) protocol. A precise volume of 30 ml of a 0.4 M glycine solution, adjusted to a pH of 1.5 using hydrochloric acid (HCl), will be added to 1.5g of all samples.

   The samples will be subjected to agitation on an orbital shaker at a speed of 250 revolutions per minute (rpm) for 2 hours, maintaining a temperature of 37°C. Subsequently, the samples will be centrifuged at a relative centrifugal force of 3000 (rcf) for a duration of 10 minutes. The resultant supernatant will be passed through a polyethersulfone (PES) filter with a pore size of 0.22 µm into a clean 50 ml centrifuge tube.

   To prepare the extracted samples for analysis, 1 ml of each sample will be diluted to a final volume of 10 ml using ultrapure deionized water. No further acidification will be performed after the dilution step. The diluted samples will be stored in a refrigerator at a temperature of 4°C until further analysis which will be performed utilising inductively coupled plasma mass spectrometry (ICP-MS) Thermo-Fisher Scientific iCAP-Q instrument manufactured by Thermo Fisher Scientific Quality Control Measures The equipment to be used will be calibrated using standard solutions and certified reference materials containing a known amount of the micronutrients being analysed before analyses will be conducted. The analytical methods used are well-established in literature for validation. The analyses will be conducted multiple times, and statistical analyses (One-way ANOVA) will be performed to determine the differences in the mean of the various foods.

ELIGIBILITY:
Inclusion Criteria:

* • Couples with a child between 6-10 years'

  * The woman is between ages 15-49 years.
  * Couples will be staying within the selected community for at least 6 months after the recruitment.

Exclusion Criteria:

* • Single parents in the study community

  * Bachelors and spinsters
  * Couples without children.
  * Married women 14 years or below and 50 years or more
  * Couples with children below or above the ages of 6-10 years.
  * Couples who fall within the inclusion criteria but have the intension of relocating from the study community within the study period.

Ages: 6 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Change in mean Nutritional Knowledge from baseline to endline | From enrollment to end of intervention at 6 months
  Nutritional Knowledge will be meansured using questionnaire. An adapted knowledge score scale (0, 1: where 0 is the least and 1 highest) will be used in scoring the participants knowledge. Participants score 1 if the answer knowledge question correctly and will score zero if they get the question wrong. There will be 11 questions on nutritional knowledge, if participants answer 9 and above questions correctly (80% and above) , they will be described as having good knowledge, 6-8 correct answers (50-70%) will be moderate knowledge while 0-5 (< 50%) correct answers will be poor knowledge. Data will be collected three times (baseline, midline and endline). The mean difference will be established based on p-value < 0.05 using repeated ANOVA
Change in mean Nutritional Attitude will be measuered from baseline to end line 6 months | From enrollment to the end of the intervention at 6 months
  A questionnaire will be used collect data on Nutritional Attitude at baseline, midline and endline. To measure change in nutritional attitude towards the consumption of green leafy vegetables, legumes and vitamin C rich fruits, two categories will be created: good attitude and poor attitude. A median score will be used to measure change in attitude based on seven (7) attitudinal questions. Participants who surpased the median score of the 7 questions will be described as having good attitude while those who score below the median will be described as having poor attidude. The mean difference will be established based on p-value < 0.05 in repeated measures using ANOVA
Change in mean will be measured for Nutritional Practice from baseline to end line at 6 months | From enrollment to the end of the intervention at 6 months
  A questionnaire will be used to measure the change in Nutritional Practice of participants. The measurement will be done using an adapted nutritional practice scale of 0 and 1, with 1 for a correct answer and 0 for a wrong answer. There will be 23 nutritional practice questions divided into 7 sections, and there will be two categorie; good or poor practice. Participants who score 16 out of 23 questions correctly (70%) and above will be classified as having good practice while those who score less than 16 out of the 23 questions correctly will be classified as having poor practice. Data will be collected at three time points: baseline, midline and endline. Mean difference will be established using repeated ANOVA and p-value < 0.05
Differences in the mean of chemical compositions of the indigenous green leafy vegetables and legumes will be measured during the study | This will be done at the end of the nutrition education intervention at 6 months
  The commonly consumed green leafy vegetables and legumes consumed by intervention group participants will be analysed in the laboratory to determine their chemical composition and iron bioaccessibity in them. The quantities of nutrients and iron bioaccessibility will be measure in mg/ 100g.One way ANOVA will be used to establish the mean differences in the vegetables and legumes at p-value < 0.005.

SECONDARY OUTCOMES:
Change in the frequency of consumption of green leafy vegetables and legumes will be measured from baseline to end line at 6 months | From enrollment to end line at 6 months
  A questionnare will be used to collect data on consumption patterns of green leafy vegetables, legumes and fruits among participants at baseline, midline and endline. There will be four options provided on the questionnaire which will include never, 1-2 times, 3-4 times, and 5-7 times per week to measure the frequency of consumption. Pearson's Chi-Square tests will be used to measure the correlation between the number of times participants consumed foods in the listed food groups per week and the food consumed.
Change in mean haemoglobin levels will be measured at baseline and endline at 6 months | At enrollment and endline at 6 months
  Haemoglobin levels (g/dL) of intervention group households (couples; father, mother and their child) will be measured at start of the intervention and at the end line of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: John Anoku, PhD, MSc, Study Chair — University of Ghana
Locations (1):
- University of Ghana, Legon, Department of Nutrition and Food Science, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underline the objectives and results of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years after publication of results
Access Criteria: IPD will be shared upon request with researchers in the field of Nutrition and Public Health who will submit data sharing agreement plan which will be reviewed by study Chair and Directors

REFERENCES:
- [Background] Zelalem, A., Endeshaw, M., Ayenew, M., Shiferaw, S., & Yirgu, R. (2017). Effect of nutrition education on pregnancy specific nutrition knowledge and healthy dietary practice among pregnant women in Addis Ababa. Clinics in Mother and Child Health, 14(3), 265.
- [Background] Yetnayet, M., Henry, C. J., Berhanu, G., Whiting, S. J., & Regassa, N. (2017). Nutrition education promoted consumption of pulse based foods among rural women of reproductive age in Sidama Zone, Southern Ethiopia. African Journal of Food, Agriculture, Nutrition and Development, 17(3), 12377-12395.
- [Background] World Health, O. (2011). Haemoglobin concentrations for the diagnosis of anaemia and assessment of severity.
- [Background] WHO. (2019). Healthy diet / World Health Organization. Regional Office for the Eastern Mediterranean. https://apps.who.int/iris/bitstream/handle/10665/325828/EMROPUB_2019_en_23536.pdf
- [Background] WHO. (2020). WHO guidance helps detect iron deficiency and protect brain development; April 2020
- [Background] Wagner MG, Rhee Y, Honrath K, Blodgett Salafia EH, Terbizan D. Nutrition education effective in increasing fruit and vegetable consumption among overweight and obese adults. Appetite. 2016 May 1;100:94-101. doi: 10.1016/j.appet.2016.02.002. Epub 2016 Feb 2. PMID 26850310
- [Background] Van Jaarsveld, P., Faber, M., Van Heerden, I., Wenhold, F., van Rensburg, W. J., & Van Averbeke, W. (2014). Nutrient content of eight African leafy vegetables and their potential contribution to dietary reference intakes. Journal of Food Composition and Analysis, 33(1), 77-84.
- [Background] Marías, Y. F., & Glasauer, P. (2014). Guidelines for assessing nutrition-related knowledge, attitudes and practices: Food and Agriculture Organization of the United Nations (FAO).
- [Background] Umeobika, U. C., Nwali, D. C., & Ekwueme, I. J. (2015). Quantitative evaluation of anti-nutritional factors in mango (Mangifera indica) fruit. Int. J. Appl. Sci. Math, 2(5), 2394-2894.
- [Background] Tuli, R. T., Rahman, M. M., Abdullah, A. T., Akhtauzzaman, M., & Islam, S. N. (2016). Phytochemicals-Tannins in some Leafy Vegetables of Bangladesh. J. Nutr, 3, 150.
- [Background] Stuetz W, Gowele V, Kinabo J, Bundala N, Mbwana H, Rybak C, Eleraky L, Lambert C, Biesalski HK. Consumption of Dark Green Leafy Vegetables Predicts Vitamin A and Iron Intake and Status among Female Small-Scale Farmers in Tanzania. Nutrients. 2019 May 7;11(5):1025. doi: 10.3390/nu11051025. PMID 31067775
- [Background] Stevens GA, Finucane MM, De-Regil LM, Paciorek CJ, Flaxman SR, Branca F, Pena-Rosas JP, Bhutta ZA, Ezzati M; Nutrition Impact Model Study Group (Anaemia). Global, regional, and national trends in haemoglobin concentration and prevalence of total and severe anaemia in children and pregnant and non-pregnant women for 1995-2011: a systematic analysis of population-representative data. Lancet Glob Health. 2013 Jul;1(1):e16-25. doi: 10.1016/S2214-109X(13)70001-9. Epub 2013 Jun 25. PMID 25103581
- [Background] Santos WPC, Ribeiro NM, Santos DCMB, Korn MGA, Lopes MV. Bioaccessibility assessment of toxic and essential elements in produced pulses, Bahia, Brazil. Food Chem. 2018 Feb 1;240:112-122. doi: 10.1016/j.foodchem.2017.07.051. Epub 2017 Jul 11. PMID 28946232
- [Background] Rosi A, Paolella G, Biasini B, Scazzina F; SINU Working Group on Nutritional Surveillance in Adolescents. Dietary habits of adolescents living in North America, Europe or Oceania: A review on fruit, vegetable and legume consumption, sodium intake, and adherence to the Mediterranean Diet. Nutr Metab Cardiovasc Dis. 2019 Jun;29(6):544-560. doi: 10.1016/j.numecd.2019.03.003. Epub 2019 Mar 14. PMID 31078365
- [Background] Rosenstock IM. Why people use health services. Milbank Mem Fund Q. 1966 Jul;44(3):Suppl:94-127. No abstract available. PMID 5967464
- [Background] Nomkong, R. F., Ejoh, R. A., Dibanda, R. F., Gabriel, M. N. J. F., & Sciences, N. (2019). Bioavailability of Iron and Related Components in Cooked Green Leafy Vegetables Consumed in Cameroon. 10(9), 1096-1111.
- [Background] Murty, P., Rao, M. V., & Bamji, M. S. (2016). Impact of enriching the diet of women and children through health and nutrition education, introduction of homestead gardens and backyard poultry in rural India. Agricultural Research, 5, 210-217.
- [Background] Lion R, Arulogun O, Titiloye M, Shaver D, Jain A, Godwin B, Sidibe M, Adejumo M, Rosseel Y, Schmidt P. The effect of the "Follow in my Green Food Steps" programme on cooking behaviours for improved iron intake: a quasi-experimental randomized community study. Int J Behav Nutr Phys Act. 2018 Aug 16;15(1):79. doi: 10.1186/s12966-018-0710-4. PMID 30115087
- [Background] Leafy green crops to improve diets on Pacific islands. Bull World Health Organ. 2018 Sep 1;96(9):595-596. doi: 10.2471/BLT.18.020918. PMID 30262939
- [Background] Holdsworth M, Pradeilles R, Tandoh A, Green M, Wanjohi M, Zotor F, Asiki G, Klomegah S, Abdul-Haq Z, Osei-Kwasi H, Akparibo R, Bricas N, Auma C, Griffiths P, Laar A. Unhealthy eating practices of city-dwelling Africans in deprived neighbourhoods: Evidence for policy action from Ghana and Kenya. Glob Food Sec. 2020 Sep;26:100452. doi: 10.1016/j.gfs.2020.100452. PMID 33324537
- [Background] Fallah F, Pourabbas A, Delpisheh A, Veisani Y, Shadnoush M. Effects of nutrition education on levels of nutritional awareness of pregnant women in Western iran. Int J Endocrinol Metab. 2013 Summer;11(3):175-8. doi: 10.5812/ijem.9122. Epub 2013 Jul 1. PMID 24348589
- [Background] de Jager I, Borgonjen-van den Berg KJ, Giller KE, Brouwer ID. Current and potential role of grain legumes on protein and micronutrient adequacy of the diet of rural Ghanaian infants and young children: using linear programming. Nutr J. 2019 Feb 21;18(1):12. doi: 10.1186/s12937-019-0435-5. PMID 30791898
- [Background] Dahanayake DN, Castillejos AG, Chodosh J, Vavvas DG. Visual restoration with KPro after face allotransplantation with a grade III phthisical eye. Digit J Ophthalmol. 2024 Jun 24;30(2):45-47. doi: 10.5693/djo.02.2024.03.003. eCollection 2024. PMID 38962671
- [Background] Coomson JB, Aryeetey R. Perception and practice of breastfeeding in public in an urban community in Accra, Ghana. Int Breastfeed J. 2018 May 18;13:18. doi: 10.1186/s13006-018-0161-1. eCollection 2018. PMID 29796057
- [Background] Bundala N, Kinabo J, Jumbe T, Bonatti M, Rybak C, Sieber S. Gaps in knowledge and practice on dietary consumption among rural farming households; a call for nutrition education training in Tanzania. Int J Food Sci Nutr. 2020 May;71(3):341-351. doi: 10.1080/09637486.2019.1655533. Epub 2019 Aug 21. PMID 31433686
- [Background] Arasaretnam, S., Kiruthika, A., & Mahendran, T. (2018). Nutritional and mineral composition of selected green leafy vegetables. Ceylon Journal of Science, 47(1), 35-41.
- [Background] Amagloh FK, Atuna RA, McBride R, Carey EE, Christides T. Nutrient and Total Polyphenol Contents of Dark Green Leafy Vegetables, and Estimation of Their Iron Bioaccessibility Using the In Vitro Digestion/Caco-2 Cell Model. Foods. 2017 Jul 22;6(7):54. doi: 10.3390/foods6070054. PMID 28737681
- [Background] Aggarwal M, Devries S, Freeman AM, Ostfeld R, Gaggin H, Taub P, Rzeszut AK, Allen K, Conti RC. The Deficit of Nutrition Education of Physicians. Am J Med. 2018 Apr;131(4):339-345. doi: 10.1016/j.amjmed.2017.11.036. Epub 2017 Dec 18. PMID 29269228
- [Background] Abu-Baker NN, Eyadat AM, Khamaiseh AM. The impact of nutrition education on knowledge, attitude, and practice regarding iron deficiency anemia among female adolescent students in Jordan. Heliyon. 2021 Feb 27;7(2):e06348. doi: 10.1016/j.heliyon.2021.e06348. eCollection 2021 Feb. PMID 33718648